CLINICAL TRIAL: NCT04710407
Title: A Phase 1, Single-center, Open-label Study to Assess the Intrapulmonary Pharmacokinetics of SPR859 by Comparing the Plasma, Epithelial Lining Fluid (ELF), and Alveolar Macrophages (AM) Concentrations Following the Oral Administration of Five Doses of SPR994 in Healthy, Nonsmoking Volunteers
Brief Title: Study to Assess the Intrapulmonary Pharmacokinetics of SPR859 by Comparing the Plasma, Epithelial Lining Fluid (ELF), and Alveolar Macrophages (AM) Concentrations Following the Oral Administration of Five Doses of SPR994 in Healthy, Nonsmoking Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Spero Therapeutics (Industry)
Collaborators: Clinartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPR994-108
Record Dates: First submitted 2021-01-04; First posted 2021-01-14 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Healthy Volunteers
Keywords: pharmacokinetics; TBPM-PI-HBr; tebipenem; alveolar macrophages (AM); epithelial lining fluid (ELF); intrapulmonary
MeSH Terms: interventions — tebipenem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TBPM-PI-HBr (Experimental): Healthy subjects meeting eligibility criteria will receive a total of five doses of TBPM-PI-HBr 600 mg orally every 8 hours.
  Interventions: Drug: TBPM-PI-HBr

INTERVENTIONS:
Drug: TBPM-PI-HBr — TBPM-PI-HBr (2 x 300mg tablets) a total of five doses
  Other Names: TBPM-PI-HBr oral capsule; SPR994

SUMMARY:
To evaluate the intrapulmonary pharmacokinetics (PK), including ELF and AM concentrations, of SPR859 (tebipenem) compared to plasma concentrations of SPR859 (tebipenem) (the active moiety in plasma of the prodrug SPR994) in nonsmoking healthy adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Adult males or female subjects, between 18 and 55 years of age (both inclusive) at the time of screening
* BMI ≥ 18.5 and ≤ 32 (kg/m2) and weight between 55.0 and 100.0 kg (both inclusive)
* Willing and able to provide written informed consent; Willing and able to comply with all study assessments and adhere to the protocol schedule
* Medically healthy without clinically significant abnormalities as assessed by the Investigator based on screening medical history, physical examination, vital signs, 12-lead ECG, hematology, biochemistry and urinalysis
* Have suitable venous access for blood sampling

Exclusion Criteria:

* History of seizure disorders
* Positive urine drug, alcohol or cotinine testing at screening or check-in (Day -1)
* Positive testing for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C antibodies (HCV);
* Positive testing for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) at screening;
* Presence of the following symptoms at screening or within 14 days prior to screening or Check-in (Day -1)

  1. Fever, chills or sweats (temperature of 38 °C / 100.4 °F or higher)
  2. Difficulty breathing
  3. Cough
  4. Sore throat
  5. New or recent loss of taste or smell
  6. Nausea, vomiting or diarrhea;
* Close contact with anyone who tested positive for SARS-CoV-2 infection within 14 days prior to screening or Check-in (Day -1);
* Electrocardiogram (ECG) with QTcF interval duration equal or greater than 450 msec for males and 470 msec for females
* Subjects who have any of the following abnormalities on laboratory values at screening or prior confinement including:

  1. White blood cell count < 3,000/mm3, hemoglobin < 11g/dL;
  2. Absolute neutrophil count <1,200/mm3, platelet count <120,000/mm3;
  3. alanine aminotransferase (ALT) and aspartate aminotransferase (AST) greater than 1.5 x the upper limit of normal (ULN) for the reference laboratory;
* History of substance abuse or alcohol abuse
* Use of tobacco/nicotine- or marijuana-containing products (including vaping products) within 12 months prior to screening;
* Known history of clinically significant hypersensitivity reaction or anaphylaxis to any medication

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-12-07 (Actual); Primary Completion 2021-03-10 (Actual); Study Completion 2021-03-10 (Actual)

PRIMARY OUTCOMES:
Plasma PK and lung penetration of SPR859 following multiple doses | Day 1 to Day 3
  Plasma PK parameters will include the area under the curve (AUC) from time zero to the last quantifiable sample (AUC0-t), AUC from time zero to end of dosing interval (AUC0-8). The AUC0-8 values for ELF and AM will be determined. The ratios of the AUC0-8 of ELF to the AUC0-8 of plasma and the AUC0-8 of AM to the AUC0-8 of plasma will be calculated.
Plasma PK and lung penetration of SPR859 following multiple doses | Day 1 to Day 3
  Plasma PK parameters will include the maximum concentration (Cmax), minimum concentration (Cmin), time to Cmax (tmax), and the terminal-phase half-life (t1/2).

SECONDARY OUTCOMES:
Safety and tolerability, including adverse events (AEs) | Day 1 to Day 10
  Frequency of adverse events by severity, seriouness, system organ class, preferred term and treatment group
Safety and tolerability, including clinically significant changes from baseline in clinical laboratory values | Day 1 to Day 10
  Change from baseline in selected laboratory assays including WBC, hemoglobin, platelet count, liver function tests (AST, ALT, AP), blood urea nitrogen (BUN), serum creatinine (Cr), and estimated Cr clearance (based on Cockcroft-Gault formula), by treatment group
Safety and tolerability, including physical examination | Day 1 to Day 10
  Change from baseline in vital signs
Safety and tolerability, including ECG | Day 1 to Day 10
  Cardiac (12-Lead ECG) will be summarized at each scheduled time point using descriptive statistics

CONTACTS AND LOCATIONS:
Overall Officials: David Baratz, MD, Principal Investigator — Pulmonary Associates
Locations (1):
- Pulmonary Associates, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rodvold KA, Gotfried MH, Gupta V, Ek A, Srivastava P, Talley A, Bruss J. Plasma and Intrapulmonary Concentrations of Tebipenem following Oral Administration of Tebipenem Pivoxil Hydrobromide to Healthy Adult Subjects. Antimicrob Agents Chemother. 2022 Jul 19;66(7):e0059022. doi: 10.1128/aac.00590-22. Epub 2022 Jun 28. PMID 35762796